CLINICAL TRIAL: NCT00360971
Title: A Randomized, Phase III, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Palifermin (NSC# 740548; IND # 6370) for the Reduction of Oral Mucositis in Patients With Locally Advanced Head and Neck Cancer Receiving Radiation Therapy With Concurrent Chemotherapy (Followed by Surgery for Selected Patients)
Brief Title: Palifermin in Lessening Oral Mucositis in Patients Undergoing Radiation Therapy and Chemotherapy for Locally Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to positive preliminary results from other palifermin studies.
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RTOG-0435; CDR0000491088
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Head and Neck Cancer; Mucositis; Pain; Radiation Toxicity
Keywords: mucositis; pain; radiation toxicity; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Pain; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck | interventions — Fibroblast Growth Factor 7; Cisplatin; Neck Dissection; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palifermin (Experimental): Concurrent radiation therapy, cisplatin, and palifermin followed by neck dissection for indicated patients.
  Interventions: Biological: palifermin; Drug: cisplatin; Procedure: neck dissection; Radiation: radiation therapy
- Placebo (Placebo Comparator): Concurrent radiation therapy, cisplatin, and placebo followed by neck dissection for indicated patients.
  Interventions: Drug: cisplatin; Other: placebo; Procedure: neck dissection; Radiation: radiation therapy

INTERVENTIONS:
Biological: palifermin — Four doses of palifermin, 180ųg/kg, administered as an i.v. bolus injection over 30-60 seconds. Starting on day -3 (Friday) prior to radiation therapy / chemotherapy and then once weekly, on days 5, 12, and 19.
  Arms: Palifermin
Drug: cisplatin — Patients will receive cisplatin (100 mg/m2) administered intravenously on days 1, 22, and 43 of the treatment course.
Other: placebo — Four doses of placebo, 180ųg/kg, administered as an i.v. bolus injection over 30-60 seconds. Starting on day -3 (Friday) prior to radiation therapy / chemotherapy and then once weekly, on days 5, 12, and 19.
  Arms: Placebo
Procedure: neck dissection — A neck dissection is required for patients with persistent nodal disease, any stage, if a palpable abnormality or worrisome radiographic abnormality persists in the neck 8-9 weeks after completion of therapy. A neck dissection is optional for patients with multiple positive lymph nodes or with lymph nodes exceeding 3 cm in diameter at pre-treatment (N2a, N2b, N3) who achieve a complete clinical and radiographic response in the neck. All patients will be assessed at approximately 8 weeks post-treatment with CT scan or MRI by the same technique used at baseline.
Radiation: radiation therapy — A radiation dose of 70 Gy with at least 66 Gy to at least 2 mucosal sites of the oral cavity/oropharynx mucosa. Radiation therapy can be given with 3D conformal (3D-CRT) or with intensity modulated RT (IMRT) techniques; however, the chosen modality must be used for the entire course of treatment.

SUMMARY:
RATIONALE: Growth factors, such as palifermin, may lessen the severity of mucositis, or mouth sores, in patients receiving radiation therapy and chemotherapy for head and neck cancer. It is not yet known whether palifermin is more effective than a placebo in lessening mucositis in patients receiving radiation therapy and chemotherapy for head and neck cancer.

PURPOSE: This randomized phase III trial is studying palifermin to see how well it works compared to a placebo in lessening oral mucositis in patients undergoing radiation therapy and chemotherapy for locally advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of palifermin vs placebo, in terms of burden of acute mucositis (defined to be 105 days [15 weeks] or less from the start of treatment), in patients with squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx undergoing concurrent radiotherapy and chemotherapy.

Secondary

* Compare incidence and time to onset of Grades 3 or 4 oral mucositis in patients treated with these regimens.
* Compare overall and progression-free survival and time to second primary in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease stage (III vs IVA or IVB), tumor site (oral cavity or oropharynx vs hypopharynx or larynx), and radiotherapy technique used on study (intensity-modulated radiotherapy [IMRT] vs 3-dimensional conformal radiotherapy [3D-CRT]). Patients are randomized to 1 of 2 treatment arms.

Mucositis, pain, and symptom burden are assessed at baseline, during radiotherapy, and post radiotherapy. Xerostomia is assessed at baseline, during radiotherapy, and several times after completion of study therapy.

After completion of study therapy, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 298 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven (from primary lesion and/or lymph nodes) diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx;
2. Patients must have at least 2 mucosal sites of the oral cavity/oropharynx mucosa assessable by visual transoral inspection that will receive at least 66 Gy;

   -2.1 Patients with tumors of the larynx or hypolarynx are eligible only if it is anticipated that the 2 index sites in the oral cavity/oropharynx mucosa will receive at least 66 Gy;
3. Patients must be able to be evaluated for the primary endpoint; therefore, patients must be able to eat at least soft solids and not require a feeding tube for nutrition or hydration at study entry.
4. Selected Stage III (excluding T1N1MO) or IVA-B (AJCC, 6th edition) at study entry, including no distant metastases, based upon the following minimum diagnostic workup:

   * 4.1 History/physical examination, including documentation of tobacco/alcohol use and current medications (including opioids/dosing), within 8 weeks prior to registration;
   * 4.2 Chest x-ray (or Chest CT scan) within 6 weeks prior to registration;
   * 4.3 MRI or CT scan with contrast of tumor site within 6 weeks prior to registration;
   * 4.4 Assessment of mucositis and xerostomia within 2 weeks prior to registration;
5. Zubrod Performance Status 0-1;
6. Age > 18;
7. Adequate bone marrow function, defined as follows:

   * 7.1 Absolute neutrophil count (ANC) > 1,800 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to registration on study
   * 7.2 Platelets > 100,000 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to registration on study
   * 7.3 Hemoglobin > 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to registration on study (Note: The use of transfusion or other intervention to achieve Hgb > 8.0 g/dl is acceptable.)
8. Adequate hepatic function with bilirubin < 1.5 mg/dl, AST or ALT < 2 x ULN within 2 weeks prior to registration;
9. Adequate renal function with serum creatinine < 1.5 mg/dl and creatinine clearance (CC) ≥ 50 ml/min within 2 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula:

   CCr male = [(140 - age) x (wt in kg)]/[(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
10. Normal serum calcium or normal corrected serum calcium within 2 weeks prior to registration; formula for corrected calcium if albumin valued is below normal range: Corrected calcium (mg/dl) = (4 - [patient's albumin (g/dl)] x 0.8) + patient's measured calcium (mg/dl);
11. Serum pregnancy test for women of childbearing potential within 2 weeks prior to registration;
12. Women of childbearing potential and male participants must practice adequate contraception.
13. Patient agrees to refrain from using all products listed in Section 9.2, "Non-permitted Supportive Therapy";
14. Patient must sign study specific informed consent prior to study entry.

Exclusion Criteria:

1. Patients with a history of prior head and neck squamous cancer are ineligible;
2. Stage IVC (AJCC, 6th edition) [Any T, Any N, M1] or distant metastases at protocol study entry; T1N1M0 patients are excluded.
3. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years;
4. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable. See Sections 1 and 3.
5. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
6. Initial surgical treatment, excluding diagnostic biopsy of the primary site or nodal sampling of neck disease; radical or modified neck dissection is not permitted.
7. Severe, active co-morbidity, defined as follows:

   * 7.1 Symptomatic and/or uncontrolled cardiac disease, New York Heart Association Classification III or IV (see Appendix II);
   * 7.2 Transmural myocardial infarction within the last 6 months;
   * 7.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * 7.4 Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
   * 7.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
   * 7.6 Patients known to be sero-positive for hepatitis B virus (HBV) or hepatitis C virus (HCV);
   * 7.7 Patients known to be sero-positive for human immunodeficiency virus (HIV) or patients with Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with HIV or AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * 7.8 A history of pancreatitis.
8. Collagen vascular disease, such as scleroderma, as this disease is thought to predispose patients to increased risk for radiation-associated toxicities;
9. Previous treatment with palifermin or other keratinocyte growth factors, such as velafermin or repifermin;
10. Prior allergic reaction or known sensitivity to any of the agents administered during dosing, including E. coli-derived products, such as Nutropin®, Neupogen®, Humulin®, Roferon®; Neumega®, Neulasta®), IntronA®, Betaseron®;
11. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David I. Rosenthal, MD, Study Chair — M.D. Anderson Cancer Center
Locations (48):
- United States (47):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Torrance Memorial Medical Center, Torrance, California
  - Solano Radiation Oncology Center, Vacaville, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Sharon Regional Cancer Care Center- Hermitage, Hermitage, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Somerset Oncology Center, Somerset, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Johnson City Medical Center Hospital, Johnson City, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
- Cross Cancer Institute at University of Alberta, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Palifermin
Started | 10 | 11
Completed | 10 (Subjects with data for planned primary analysis are considered to have completed the study.) | 11 (Subjects with data for planned primary analysis are considered to have completed the study.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Palifermin | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Full Range); unit: years] | 52 [35 to 82] | 55 [48 to 67] | 55 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Duration of Oral Mucositis as Measured in Terms of Days
Description: Duration in days of World Heath Organization (WHO) Grades 3 and 4 oral mucositis during the acute period (defined to be 105 days [15 weeks] or less from the start of treatment); duration is calculated from the onset of a Grade 3 or 4 oral mucositis to the day when an oral mucositis of ≤ Grade 2 is reported after the last oral mucositis of Grade 3 or 4. Patients with grade 0-2 mucositis have a duration of 0.
  This study required 298 patients to detect via two-sided t-test a reduction of mean duration of at least 9 days from 29 days (standard deviation = 23 days) on the placebo arm with 90% power and alpha = 0.05.
  Statistical testing was not done due to the small sample size.
Time Frame: Twice-weekly from start of treatment up to 15 weeks after the start of treatment.
Population: All eligible patients.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 10 | 11
Days | 32 (24) | 13 (23)

2. Secondary Outcome: Number of Patients With Grade 3 or 4 Mucositis as Measured by the World Heath Organization (WHO) Scale
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: Twice-weekly from start of treatment up to 15 weeks after the start of treatment.
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 10 | 11
Participants | 8 | 4

3. Secondary Outcome: Time to Onset of Grade 3 or 4 Oral Mucositis as Measured by the World Heath Organization (WHO) Scale
Description: as for outcome 2
Time Frame: Twice-weekly from start of treatment up to 15 weeks after the start of treatment.
Population: All randomized patients
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 10 | 11
days | 48 (10) | 41 (6)

4. Secondary Outcome: Overall Survival
Description: An event is death from any cause. Overall survival was not calculated due to the limited number of events. Number of patients with an event is reported.
Time Frame: From randomization to maximum follow-up at time of analysis of 21 months
Population: Randomized patients who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 8 | 11
Participants | 2 | 0

5. Secondary Outcome: Progression-free Survival
Description: An event is defined as the first occurrence of local, regional, distant disease. Progression-free survival is calculated at the time from registration to the death of progression, death in the absence of progression, or last follow-up. Progression-free survival was not calculated due to the limited number of events. Number of patients with an event is reported.
Time Frame: From randomization to maximum follow-up at time of analysis of 21 months
Population: Randomized patients who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 8 | 11
Participants | 2 | 0

6. Secondary Outcome: Time to Second Primary Tumor
Description: An event is occurrence of a second primary other than basal cell. Time to second primary tumor was not calculated because there were no events. Number of patients with an event is reported.
Time Frame: From randomization to maximum follow-up at time of analysis of 21 months
Population: Randomized patients who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given SAE (serious adverse event) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE). Mucositis was collected separately from other AE's using the World Health Organization (WHO) grading criteria.
Arm/Group | Placebo | Palifermin
Serious Adverse Events (participants affected / at risk) | 8/10 | 5/11
Other Adverse Events (participants affected / at risk) | 9/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Palifermin (N=11)
Mucositis (Gastrointestinal disorders) | 8 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Appendix (Infections and infestations) | 1 | 0
Metabolic/laboratory - Other: (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 1 | 0
Renal/genitourinary - Other: (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular - Other: (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Palifermin (N=11)
Hemoglobin (Blood and lymphatic system disorders) | 4 | 5
Hearing impaired (Ear and labyrinth disorders) | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 2
Endocrine - Other: (Endocrine disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 2 | 7
Caecitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhoea NOS (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 7 | 9
Dysphagia (Gastrointestinal disorders) | 3 | 6
Esophageal stenosis acquired (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other: (Gastrointestinal disorders) | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4
Oral pain (Gastrointestinal disorders) | 2 | 2
Oseophagitis NOS (Gastrointestinal disorders) | 2 | 1
Salivary gland disorder NOS (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 3
Edema: head and neck: (General disorders) | 3 | 0
Fatigue (General disorders) | 5 | 2
Pyrexia (General disorders) | 0 | 1
Infection - Other: (Infections and infestations) | 2 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Mucosa (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Pharynx (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Neck NOS (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Upper aerodigestive NOS (Infections and infestations) | 0 | 1
Infection with unknown ANC: Oral cavity-gums (gingivitis) (Infections and infestations) | 1 | 0
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 2 | 2
Ecchymosis (Injury, poisoning and procedural complications) | 1 | 0
Radiation recall syndrome (Injury, poisoning and procedural complications) | 2 | 2
Alanine aminotransferase increased (Investigations) | 3 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 2
Coagulopathy (Investigations) | 0 | 1
Leukopenia NOS (Investigations) | 5 | 3
Lymphopenia (Investigations) | 1 | 1
Metabolic/laboratory - Other: (Investigations) | 2 | 2
Neutrophil count (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 5 | 7
Anorexia (Metabolism and nutrition disorders) | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibrosis-deep connective tissue: (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 1 | 0
Laryngeal nerve dysfunction: (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Myelitis NOS (Nervous system disorders) | 1 | 0
Neuralgia NOS (Nervous system disorders) | 1 | 0
Neurology - Other: (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 0
Trigeminal nerve disorder NOS (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study terminated early with 21 subjects accrued out of 298 planned, therefore no statistical testing was performed. The termination was decided due to positive preliminary results from other palifermin studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.